CLINICAL TRIAL: NCT02102984
Title: Covered Versus Uncovered Metal Stents for Biliary Malignancies - A Randomized Controlled Trial
Brief Title: Covered Versus Uncovered Biliary Stents for Biliary Malignancies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nuovo Ospedale Civile S.Agostino Estense (Other)
Responsible Party: Principal Investigator, Rita Conigliaro, MD, Chief - Endoscopy Unit, Nuovo Ospedale Civile S.Agostino Estense
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 242/13
Record Dates: First submitted 2014-03-26; First posted 2014-04-03 (Estimated); Last update posted 2016-03-30 (Estimated); Status verified 2016-03

CONDITIONS: Biliary Tract Cancer
Keywords: distal malignancy of the extra-hepatic biliary tract; metallic biliary stents; covered biliary stents; uncovered biliary stents
MeSH Terms: conditions — Biliary Tract Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- covered stents (Active Comparator): endoscopic placement of covered biliary stents
  Interventions: Device: covered biliary stents
- uncovered biliary stents (Active Comparator): endoscopic placement of uncovered biliary stents
  Interventions: Device: uncovered biliary stents

INTERVENTIONS:
Device: covered biliary stents — endoscopic placement of covered biliary stents
  Other Names: Taewoong Medical NITI-S Covered
  Arms: covered stents
Device: uncovered biliary stents — endoscopic placement of uncovered biliary stents
  Other Names: Taewoong Medical NITI-S Uncovered
  Arms: uncovered biliary stents

SUMMARY:
Patency duration of covered metal stents as compared with uncovered metal stents in the management of malignant strictures of the extra-hepatic biliary tree.

DETAILED DESCRIPTION:
Consecutive patients with malignant strictures of the extra-hepatic biliary tree considered unfit for surgical excision Placement of covered or uncovered metal stents in patients with and without gallbladder on the basis of a computer-generated randomization list Evaluation of clinical outcome, survival, complications, and quality of life. Evaluation of the cost and efficacy of the two types of metal stents.

ELIGIBILITY:
Inclusion Criteria:

* adult patients with symptomatic malignant obstruction of the extra-hepatic biliary tree
* not eligible for surgical intervention
* able to provide informed consent

Exclusion Criteria:

* benign biliary obstruction
* previous surgery of the biliary tract
* life expectancy < 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2014-04; Primary Completion 2015-09 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Relief of malignant biliary obstruction | six months
  Clinical assessment

SECONDARY OUTCOMES:
cost/effecacy | 6 months
  cost and effectiveness of covered versus uncovered biliary stents

OTHER OUTCOMES:
gallbladder in situ | 6 months
  Acute cholecystitis could affect the clinical outcome of patients when a covered stent is used

CONTACTS AND LOCATIONS:
Overall Officials: Rita Conigliaro, MD, Principal Investigator — Digestive Endoscopy Unit-NOCSAE- Modena
Locations (1):
- NOCSAE - Viale Giardini 1355, Modena, Italy

REFERENCES:
- [Background] Isayama H, Nakai Y, Kogure H, Yamamoto N, Koike K. Biliary self-expandable metallic stent for unresectable malignant distal biliary obstruction: which is better: covered or uncovered? Dig Endosc. 2013 May;25 Suppl 2:71-4. doi: 10.1111/den.12078. PMID 23617653
- [Derived] Conio M, Mangiavillano B, Caruso A, Filiberti RA, Baron TH, De Luca L, Signorelli S, Crespi M, Marini M, Ravelli P, Conigliaro R, De Ceglie A. Covered versus uncovered self-expandable metal stent for palliation of primary malignant extrahepatic biliary strictures: a randomized multicenter study. Gastrointest Endosc. 2018 Aug;88(2):283-291.e3. doi: 10.1016/j.gie.2018.03.029. Epub 2018 Apr 11. PMID 29653120